CLINICAL TRIAL: NCT02427490
Title: A Problem-Solving Intervention for Family Caregivers in Palliative Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Karla Washington, Principal Investigator, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2002215
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Palliative Care; Caregivers; Medical Oncology
Keywords: Palliative Care; Caregivers; Medical Oncology
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unenhanced Monitoring (Active Comparator): Family caregivers of cancer patients receiving outpatient palliative care will complete standardized questionnaires at the time of study enrollment and two, four, and eight weeks after study enrollment.
  Interventions: Other: Unenhanced Monitoring
- Problem-Solving Intervention (Experimental): Family caregivers of cancer patients receiving outpatient palliative care will use videoconferencing tools to participate in three problem-solving sessions with a member of the research team.
  Interventions: Behavioral: Problem-Solving Intervention; Other: Unenhanced Monitoring

INTERVENTIONS:
Behavioral: Problem-Solving Intervention — The problem-solving approach that will be taught in the problem-solving intervention is based on the ADAPT model, which encourages participants to follow five steps when solving problems: focus on adopting a positive attitude to problem-solving, define the problem and set goals, generate a list of alternative solutions to the problem, predict consequences of the alternative solutions, and try implementing the most promising solution from among the list of alternatives. The problem-solving intervention will be delivered by a trained interventionist in three structured sessions using videoconferencing tools.
  Other Names: Problem-Solving Intervention for Family Caregivers
  Arms: Problem-Solving Intervention
Other: Unenhanced Monitoring — Study participant completes standardized questionnaires upon study enrollment and at two, four, and eight weeks after study enrollment.
  Other Names: Unenhanced Monitoring of Behavioral Health Outcomes

SUMMARY:
In congruence with the National Cancer Institute's commitment to supporting families of individuals with cancer across the full disease trajectory, the investigators seek to examine the feasibility of a technologically-mediated problem-solving intervention designed to improve the quality of life and decrease the psychological distress of family caregivers of cancer patients receiving outpatient palliative care. Investigators involved in this mixed methods pilot study will collect and analyze both quantitative and qualitative data, which will subsequently inform a large-scale randomized clinical trial of the problem-solving intervention.

DETAILED DESCRIPTION:
Palliative oncology providers are ideally situated to improve the cancer journey for the millions of family members and friends who are vital to the care of seriously ill patients. In recent decades, the primary setting for cancer care has shifted from the hospital inpatient unit to the outpatient clinic, leaving family caregivers responsible for providing the majority of patient care in the home, often with little support or preparation. The numerous stressors associated with family caregiving often give rise to caregiver anxiety, depression, fatigue, neglect of self-care and, for particularly strained caregivers, psychological symptoms that mirror those experienced by trauma survivors. In congruence with the National Cancer Institute's commitment to supporting families of individuals with cancer across the full disease trajectory, the investigators seek to examine the feasibility of a technologically-mediated problem-solving intervention designed to improve the quality of life and decrease the psychological distress of family caregivers of cancer patients receiving outpatient palliative care. Specifically, the investigators aim to 1) examine the feasibility of the intervention relative to recruitment, randomization, retention, and fidelity to core intervention components; 2) investigate the impact of the intervention on family caregiver anxiety, depression, and quality of life; and 3) explore the benefits and challenges associated with the intervention from the perspective of participants. To accomplish these aims, investigators will recruit and randomly assign 82 family caregivers of cancer patients receiving outpatient palliative care into two groups (usual care and intervention) and collect quantitative and qualitative data, which will be analyzed to inform a future large-scale randomized clinical trial of the problem-solving intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* access to an Internet-connected device that will support videoconferencing software

Exclusion Criteria:

* Younger than 18 years of age,
* lack of access to an Internet-connected device that will support videoconferencing software

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Change in anxiety (as measured by the Generalized Anxiety Disorder Form - 7) | Upon study enrollment, two weeks, four weeks, eight weeks
  Family caregivers indicate the frequency with which they experience seven different symptoms of anxiety (7 items); higher scores reflect higher anxiety severity.

SECONDARY OUTCOMES:
Change in depression (as measured by the Patient Health Questionnaire - 9) | Upon study enrollment, two weeks, four weeks, eight weeks
  Family caregivers indicate the frequency with which they experience nine different symptoms of depression (9 items); higher scores reflect higher depression severity.
Change in problem-solving approach (as measured by the Problem-Solving Inventory) | Upon study enrollment, two weeks, four weeks, eight weeks
  Family caregivers indicate the extent to which different statements describing approaches to problem-solving apply to them (25 items).
Change in quality of life (as measured by the Caregiver Quality of Life Index - Revised) | Upon study enrollment, two weeks, four weeks, eight weeks
  Family caregivers complete four items rating their physical, emotional, social, and financial quality of life on a scale of 0-10.

OTHER OUTCOMES:
Change in caregiving problems and intensity | Upon study enrollment, two weeks, four weeks, eight weeks
  Family caregivers select three problems and rate their corresponding distress using a scale of 0-3 where 0 = problem is not at all distressful and 3 = problem is very distressful (3 items).

CONTACTS AND LOCATIONS:
Overall Officials: Karla Washington, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Ambulatory Palliative Care Clinic, Columbia, Missouri, United States

REFERENCES:
- [Derived] Benson JJ, Washington KT, Landon OJ, Chakurian DE, Demiris G, Parker Oliver D. When Family Life Contributes to Cancer Caregiver Burden in Palliative Care. J Fam Nurs. 2023 Aug;29(3):275-287. doi: 10.1177/10748407231167545. Epub 2023 May 16. PMID 37190779
- [Derived] Washington KT, Benson JJ, Chakurian DE, Popejoy LL, Demiris G, Rolbiecki AJ, Oliver DP. Comfort Needs of Cancer Family Caregivers in Outpatient Palliative Care. J Hosp Palliat Nurs. 2021 Jun 1;23(3):221-228. doi: 10.1097/NJH.0000000000000744. PMID 33605647
- [Derived] Washington KT, Craig KW, Parker Oliver D, Ruggeri JS, Brunk SR, Goldstein AK, Demiris G. Family caregivers' perspectives on communication with cancer care providers. J Psychosoc Oncol. 2019 Nov-Dec;37(6):777-790. doi: 10.1080/07347332.2019.1624674. Epub 2019 Jun 16. PMID 31204604